CLINICAL TRIAL: NCT03294616
Title: Transcutaneous Electroacupuncture for Gastric Complications of Scleroderma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00089514
Record Dates: First submitted 2017-08-18; First posted 2017-09-27 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Scleroderma; Gastroparesis
Keywords: transcutaneous electroacupuncture
MeSH Terms: conditions — Scleroderma, Diffuse; Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- scleroderma patients-0 (Experimental): for acute study: The experiment in patients will be performed in 4 randomized sessions on separate days (at least 3 days apart): one control session with sham-TEA and 3 TEA sessions at various parameters. TEA will be applied on both acupoints ST36 and PC6; the following sets of parameters will be tested for TEA at ST36: A) standard parameters: the set used in the previous SSc study: 25 Hz, 0.3ms, 2s-on and 3s-off; B) same as A but pulse width of 0.6ms; C) same as B but 0.1s-on and 0.4s-off. For TEA at PC6, 25 Hz will be replaced by 100Hz because TEA at PC6 is used to treat symptoms and 100Hz is believed to be better than 25Hz. The patient will be fasted overnight, and the test will last 2 hours (1 hour fasting and 1 hour postprandial).
  Interventions: Device: transcutaneous electroacupuncture
- scleroderma patient-1 (Experimental): for chronic study: 2 weeks of Sham transcutaneous electroacupuncture treatment, 2 weeks of wash out, 2 weeks of transcutaneous electroacupuncture/Sham transcutaneous electroacupuncture treatment. Best parameter gained from acute study will be used.
  Interventions: Device: transcutaneous electroacupuncture
- scleroderma patients-2 (Experimental): for chronic study: 2 weeks of transcutaneous electroacupuncture treatment, 2 weeks of wash out, 2 weeks of transcutaneous electroacupuncture/Sham transcutaneous electroacupuncture treatment. Best parameter gained from acute study will be used.
  Interventions: Device: transcutaneous electroacupuncture

INTERVENTIONS:
Device: transcutaneous electroacupuncture — Weak electrical current will be generated by the device and delivered via skin surface electrodes to acupuncture points related to gastrointestinal functions
  Other Names: TEA

SUMMARY:
An innovative method of needleless transcutaneous electroacupuncture (TEA) using a newly developed watch-size stimulator is proposed. Weak electrical current will be delivered via skin surface electrodes to acupuncture points related to gastrointestinal functions. The stimulator can be attached to the skin near the acupuncture points and therefore daily activity of the patient does not need to be altered. Two experiments are designed to prove the feasibility of the proposed therapy for gastric complications of Scleroderma .

ELIGIBILITY:
Inclusion Criteria:

* No any systemic diseases;
* no scleroderma; no history of gastrointestinal surgery;
* no dyspeptic symptoms during the past 2 weeks;
* not taking any medications except contraceptives during the past 2 weeks;
* age 18 and older.

Exclusion Criteria:

* History of any systemic diseases or surgeries;
* allergic to adhesives; pregnancy;
* unable to sign the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 1 day
  On the first visit; The validated UCLA SCTC GIT2.0 ("University of California at Los Angeles Scleroderma Clinical Trials Consortium Gastro-Intestinal Tract Instrument version 2.0") for SSc will be the primary outcome measurement; it includes 7 categories: reflux, distention and bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 28 days
  On the second visit; The validated "University of California at Los Angeles Scleroderma Clinical Trials Consortium Gastro-Intestinal Tract Instrument version 2.0" (UCLA SCTC GIT2.0) for SSc will be the primary outcome measurement; it includes 7 categories: reflux, distention and bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 42 days
  On the third visit; The validated UCLA SCTC GIT2.0 ("University of California at Los Angeles Scleroderma Clinical Trials Consortium Gastro-Intestinal Tract Instrument version 2.0") for SSc will be the primary outcome measurement; it includes 7 categories: reflux, distention and bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 70 days
  The validated UCLA SCTC GIT2.0 ("University of California at Los Angeles Scleroderma Clinical Trials Consortium Gastro-Intestinal Tract Instrument version 2.0") for SSc will be the primary outcome measurement; it includes 7 categories: reflux, distention and bloating, fecal soilage, diarrhea, social functioning, emotional well-being and constipation
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 1 day
  Scleroderma Health Assessment Questionnaire will be used to assess SSc symptoms
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 28 days
  Scleroderma Health Assessment Questionnaire will be used to assess SSc symptoms
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 42 days
  Scleroderma Health Assessment Questionnaire will be used to assess SSc symptoms
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 70 days
  Scleroderma Health Assessment Questionnaire will be used to assess SSc symptoms
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 1 day
  SF-36 questionnaire will be used to assess general quality of life
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 28 days
  SF-36 questionnaire will be used to assess general quality of life
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 42 days
  SF-36 questionnaire will be used to assess general quality of life
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 70 days
  SF-36 questionnaire will be used to assess general quality of life
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 1 day
  a validated method including 9 symptoms will be used to assess GI symptoms
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 28 days
  a validated method including 9 symptoms will be used to assess GI symptoms
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 42 days
  a validated method including 9 symptoms will be used to assess GI symptoms
effect of TEA on symptoms in Systemic Sclerosis (SSc) patients | 70 days
  a validated method including 9 symptoms will be used to assess GI symptoms

SECONDARY OUTCOMES:
effects of TEA on gastric motility | 1 week
  visit 1 in acute phase; gastric slow waves recording
effects of TEA on gastric motility | 2 weeks
  visit 2 in acute phase; gastric slow waves recording
effects of TEA on gastric motility | 3 weeks
  visit 3 in acute phase; gastric slow waves recording
effects of TEA on gastric motility | 4 weeks
  visit 4 in acute phase; gastric slow waves recording
effects of TEA on autonomic function | 1 week
  visit 1 in acute phase; heart rate variability recording
effects of TEA on autonomic function | 2 weeks
  visit 2 in acute phase; heart rate variability recording
effects of TEA on autonomic function | 3 weeks
  visit 3 in acute phase; heart rate variability recording
effects of TEA on autonomic function | 4 weeks
  visit 4 in acute phase; heart rate variability recording
effects of TEA on gastric motility | 1 day
  visit 1 in chronic phase; gastric slow waves recording
effects of TEA on gastric motility | 28 days
  visit 2 in chronic phase; gastric slow waves recording
effects of TEA on gastric motility | 42 days
  visit 3 in chronic phase; gastric slow waves recording
effects of TEA on gastric motility | 70 days
  visit 4 in chronic phase; gastric slow waves recording
effects of TEA on gastric motility | 1 day
  visit 1 in chronic phase; breath test will be used to assess gastric emptying
effects of TEA on gastric motility | 28 days
  visit 2 in chronic phase; breath test will be used to assess gastric emptying
effects of TEA on gastric motility | 42 days
  visit 3 in chronic phase; breath test will be used to assess gastric emptying
effects of TEA on gastric motility | 70 days
  visit 4 in chronic phase; breath test will be used to assess gastric emptying
effects of TEA on autonomic function | 1 day
  visit 1 in chronic phase; heart rate variability recording
effects of TEA on autonomic function | 28 days
  visit 2 in chronic phase; heart rate variability recording
effects of TEA on autonomic function | 42 days
  visit 3 in chronic phase; heart rate variability recording
effects of TEA on autonomic function | 70 days
  visit 4 in chronic phase; heart rate variability recording
effects of TEA on autonomic function | 1 day
  visit 1 in chronic phase; Composite Autonomic Symptoms Score (COMPASS) 31 survey will be used to assess autonomic function
effects of TEA on autonomic function | 28 days
  visit 2 in chronic phase; Composite Autonomic Symptoms Score (COMPASS) 31 survey will be used to assess autonomic function
effects of TEA on autonomic function | 42 days
  visit 3 in chronic phase; Composite Autonomic Symptoms Score (COMPASS) 31 survey will be used to assess autonomic function
effects of TEA on autonomic function | 70 days
  visit 1 in chronic phase; Composite Autonomic Symptoms Score (COMPASS) 31 survey visit 4 in chronic phase; will be used to assess autonomic function
effects of TEA on autonomic function | 1 day
  baseline before the study; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 28 days
  baseline before the study; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 42 days
  baseline before the study; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 70 days
  baseline before the study; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 1 day
  30 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 28 days
  30 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 42 days
  30 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 70 days
  30 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 1 day
  60 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 28 days
  60 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 42 days
  60 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 70 days
  60 minutes after the testing meal; NE (indication of sympathetic activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 1 day
  baseline before the study; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 28 days
  baseline before the study; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 42 days
  baseline before the study; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 70 days
  baseline before the study; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 1 day
  30 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 28 days
  30 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 42 days
  30 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 70 days
  30 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 1 day
  60 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 28 days
  60 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 42 days
  60 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on autonomic function | 70 days
  60 minutes after the testing meal; pancreatic polypeptide (PP, indication of vagal activity) will be assessed using ELISA autonomic function.
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  baseline before the study; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  baseline before the study; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  baseline before the study; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  baseline before the study; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  30 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  30 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  30 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  30 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  60 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  60 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  60 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  60 minutes after the testing meal; vasoactive intestinal peptide (VIP)
effects of TEA on GI hormones and inflammatory cytokine | day 1
  baseline before the study; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  baseline before the study; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  baseline before the study; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  baseline before the study; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  30 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  30 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  30 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  30 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  60 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  60 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  60 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  60 minutes after the testing meal; interleukin-10 (IL-10)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  baseline before the study; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  baseline before the study; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  baseline before the study; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  baseline before the study; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  30 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  30 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  30 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  30 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  60 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  60 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  60 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  60 minutes after the testing meal; interferon α(IFNα)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  baseline before the study; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  baseline before the study; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  baseline before the study; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  baseline before the study; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  30 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  30 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  30 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  30 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  60 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  60 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  60 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  60 minutes after the testing meal; interleukin-1 beta (IL-1β)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  baseline before the study; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  baseline before the study; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  baseline before the study; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  baseline before the study; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  30 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  30 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  30 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  30 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  60 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  60 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  60 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  60 minutes after the testing meal; interleukin-6 (IL-6)
effects of TEA on GI hormones and inflammatory cytokine | day 1
  baseline before the study; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  baseline before the study; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  baseline before the study; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  baseline before the study; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  30 minutes after the testing meal; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  30 minutes after the testing meal; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  30 minutes after the testing meal; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  30 minutes after the testing meal; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 1 day
  60 minutes after the testing meal; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 28 days
  60 minutes after the testing meal; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 42 days
  60 minutes after the testing meal; tumor necrosis factor alpha(TNFα)
effects of TEA on GI hormones and inflammatory cytokine | 70 days
  60 minutes after the testing meal; tumor necrosis factor alpha(TNFα)

CONTACTS AND LOCATIONS:
Overall Officials: Jiande Chen, Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
haven't decided yet.